CLINICAL TRIAL: NCT00077649
Title: Randomized, Multicenter, Double-blind, Phase IV Pilot Study Evaluating the Effect of PEGASYS Doses of 180 ug or 270 ug in Combination With Copegus Doses of 1200 mg or 1600 mg on Viral Kinetics, Virological Response, Pharmacokinetics, and Safety in Interferon-naïve Patients With Chronic Hepatitis C Genotype 1 Virus Infection of High Viral Titer and Body Weight Greater Than 85 kg
Brief Title: A Study of PEGASYS (Peginterferon Alfa-2a (40KD)) in Combination With COPEGUS (Ribavirin) in Interferon-Naive Patients With Chronic Hepatitis C Infection (CHC).
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NV17318
Record Dates: First submitted 2004-02-10; First posted 2004-02-13 (Estimated); Results first posted 2016-04-18 (Estimated); Last update posted 2016-04-18 (Estimated); Status verified 2016-03

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — Ribavirin; peginterferon alfa-2a

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- PEG-IFN Alfa-2a 180 μg +Ribavirin 1200 mg (Active Comparator): Participants received 180 μg of PEG-IFN [peginterferon] alfa-2a in 1 mL solution administered [subcutaneously] sc, once weekly + 1200 mg of ribavirin (200 mg/tablet) + ribavirin placebo (2 tablets) administered [orally ] po daily in split doses for 48 weeks
  Interventions: Drug: ribavirin [Copegus]; Drug: peginterferon alfa-2a (PEG-IFN alfa-2a) [Pegasys]
- PEG-IFN Alfa-2a 180 μg + Ribavirin 1600 mg (Experimental): Participants received 180 μg of PEG-IFN [peginterferon] alfa-2a in 1 mL solution administered [subcutaneously] sc, once weekly + 1200 mg of ribavirin (200 mg/tablet) + ribavirin placebo (2 tablets) administered [orally ] po daily in split doses for 48 weeks
  Interventions: Drug: ribavirin [Copegus]; Drug: peginterferon alfa-2a (PEG-IFN alfa-2a) [Pegasys]
- PEG-IFN Alfa-2a 270 μg + Ribavirin 1200 mg (Experimental): Participants received 270 μg of PEG-IFN alfa-2a in 1-mL solution administered sc once weekly + 1200 mg of ribavirin (200 mg/tablet) + ribavirin placebo (2 tablets) administered po daily in split doses for 48 weeks
  Interventions: Drug: ribavirin [Copegus]; Drug: peginterferon alfa-2a (PEG-IFN alfa-2a) [Pegasys]
- PEG-IFN Alfa-2a 270 μg + Ribavirin 1600 mg (Experimental): Participants received 270 μg of PEG-IFN alfa-2a in 1-mL solution administered sc once weekly + 1600 mg of ribavirin (200 mg/tablet) administered po daily in split doses for 48 weeks.
  Interventions: Drug: ribavirin [Copegus]; Drug: peginterferon alfa-2a (PEG-IFN alfa-2a) [Pegasys]

INTERVENTIONS:
Drug: ribavirin [Copegus] — 600mg po bid for 48 weeks
  Arms: PEG-IFN Alfa-2a 180 μg +Ribavirin 1200 mg; PEG-IFN Alfa-2a 270 μg + Ribavirin 1200 mg
Drug: ribavirin [Copegus] — 800mg po bid for 48 weeks
  Arms: PEG-IFN Alfa-2a 180 μg + Ribavirin 1600 mg; PEG-IFN Alfa-2a 270 μg + Ribavirin 1600 mg
Drug: peginterferon alfa-2a (PEG-IFN alfa-2a) [Pegasys] — 180 micrograms sc weekly for 48 weeks
  Arms: PEG-IFN Alfa-2a 180 μg + Ribavirin 1600 mg; PEG-IFN Alfa-2a 180 μg +Ribavirin 1200 mg
Drug: peginterferon alfa-2a (PEG-IFN alfa-2a) [Pegasys] — 270 micrograms sc weekly for 48 weeks
  Arms: PEG-IFN Alfa-2a 270 μg + Ribavirin 1200 mg; PEG-IFN Alfa-2a 270 μg + Ribavirin 1600 mg

SUMMARY:
The effects of treatment with different doses of PEGASYS in combination with different doses of ribavirin will be evaluated in patients with CHC genotype 1 who have a high viral titer, body weight greater than 85kg (187lbs) and no prior treatment with interferon. The anticipated time on study treatment is 3-12 months and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients >=18 years of age;
* body weight >85kg (187lbs);
* CHC (genotype 1);
* liver biopsy (in <24 calendar months of first dose), with results consistent with CHC infection;
* use of 2 forms of contraception during study and 6 months after the study in both men and women.

Exclusion Criteria:

* women who are pregnant or breastfeeding;
* male partners of women who are pregnant;
* conditions associated with decompensated liver disease;
* other forms of liver disease, including liver cancer;
* human immunodeficiency virus infection;
* previous treatment with an interferon, ribavirin, viramidine, levovirin or amantadine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2004-01; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (24):
- United States (23):
  - La Jolla, California
  - Long Beach, California
  - San Diego, California
  - Farmington, Connecticut
  - Bradenton, Florida
  - Gainesville, Florida
  - Jacksonville, Florida
  - Wellington, Florida
  - Honolulu, Hawaii
  - Chicago, Illinois
  - Iowa City, Iowa
  - Boston, Massachusetts
  - St Louis, Missouri
  - Manhasset, New York
  - Chapel Hill, North Carolina
  - Statesville, North Carolina
  - Cincinnati, Ohio
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Houston, Texas
  - Salt Lake City, Utah
  - Charlottesville, Virginia
  - Richmond, Virginia
- Santurce, Puerto Rico

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 188 participants were enrolled in the study which was conducted at 23 centers in the United States from 13 January 2004 to 06 December 2005
Pre-assignment Details: Number of participants who completed and did not complete the 48 weeks of treatment are presented in the table .
Groups:
- PEG-IFN Alfa-2a 180 mcg +Ribavirin 1200 mg: Participants received 180 micrograms (mcg) of PEG-IFN [peginterferon] alfa-2a in 1 milliliter (mL) solution administered subcutaneously (SC), once weekly + 1200 milligrams (mg) of ribavirin (200 mg/tablet) + ribavirin placebo (2 tablets) administered [orally ] po daily in split doses for 48 weeks
- PEG-IFN Alfa-2a 180 mcg + Ribavirin 1600 mg: Participants received 180 mcg of PEG-IFN alfa-2a in 1-mL solution administered sc once weekly + 1600 mg of ribavirin (200 mg/tablet) administered po daily in split doses for 48 weeks.
- PEG-IFN Alfa-2a 270 mcg + Ribavirin 1200 mg: Participants received 270 mcg of PEG-IFN alfa-2a in 1-mL solution administered sc once weekly + 1200 mg of ribavirin (200 mg/tablet) + ribavirin placebo (2 tablets) administered po daily in split doses for 48 weeks
- PEG-IFN Alfa-2a 270 mcg + Ribavirin 1600 mg: Participants received 270 mcg of PEG-IFN alfa-2a in 1-mL solution administered sc once weekly + 1600 mg of ribavirin (200 mg/tablet) administered po daily in split doses for 48 weeks.
Period: Overall Study
Arm/Group | PEG-IFN Alfa-2a 180 mcg +Ribavirin 1200 mg | PEG-IFN Alfa-2a 180 mcg + Ribavirin 1600 mg | PEG-IFN Alfa-2a 270 mcg + Ribavirin 1200 mg | PEG-IFN Alfa-2a 270 mcg + Ribavirin 1600 mg
Started | 47 | 47 | 47 | 47
Completed 24 Weeks of Follow-up | 36 | 40 | 36 | 31
Completed | 33 | 38 | 32 | 30
Not Completed | 14 | 9 | 15 | 17
Not completed — Adverse Event | 5 | 1 | 7 | 9
Not completed — Lack of Efficacy | 5 | 3 | 3 | 2
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 2
Not completed — Lost to Follow-up | 2 | 2 | 3 | 2
Not completed — Abnormality of Laboratory Test | 1 | 2 | 1 | 2
Not completed — Randomized but never dosed | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The ITT [intent to treat] population which consisted of all participants who were randomized and received at least one dose of either of the study medication
Groups:
- PEG-IFN Alfa-2a 180 mcg+ Ribavirin 1200 mg: Participants received 180 mcg of PEG-IFN alfa-2a in 1 mL solution administered sc, once weekly + 1200 mg of ribavirin (200 mg/tablet) + ribavirin placebo (2 tablets) administered [orally ] po daily in split doses for 48 weeks.
- Total: Total of all reporting groups
Arm/Group | PEG-IFN Alfa-2a 180 mcg+ Ribavirin 1200 mg | PEG-IFN Alfa-2a 180 mcg + Ribavirin 1600 mg | PEG-IFN Alfa-2a 270 mcg + Ribavirin 1200 mg | PEG-IFN Alfa-2a 270 mcg + Ribavirin 1600 mg | Total
Number analyzed (Participants) | 47 | 47 | 47 | 47 | 188
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.2 (7.48) | 49.6 (8.46) | 47.1 (6.37) | 48.5 (6.78) | 48.1 (7.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 6 | 12 | 10 | 37
  Male | 38 | 41 | 35 | 37 | 151

OUTCOME MEASURES:

1. Primary Outcome: HCV RNA Profile During The First 24 Weeks
Description: Viral loads (quantitative HCV RNA) collected during the initial 24 weeks were first logarithmically (based 10) transformed. Results falling below the assay sensitivity level were set to the assay sensitivity level before the analyses. Thus, a qualitative HCV RNA negative result was set to 50 IU/mL (or 100 copies/mL). A qualitative HCV RNA positive result along with an unquantifiable HCV RNA result from the quantitative assay corresponded to a numeric HCV RNA result of 600 IU/mL (or 1000 copies/mL).
Time Frame: Baseline (Day 1), At 72 hour (h), Week (W)-1, 2, 4, 12, 24
Population: The ITT population consisted of all participants who were randomized and received at least one dose of either of the study medication.
Measure: Mean (Standard Deviation); unit: log 10 copies/mL
Groups:
- PEG-IFN Alfa-2a 180 mcg + Ribavirin 1200 mg: Participants received 180 mcg of PEG-IFN alfa-2a in 1 mL solution administered sc, once weekly + 1200 mg of ribavirin (200 mg/tablet) + ribavirin placebo (2 tablets) administered po daily in split doses for 48 weeks
Arm/Group | PEG-IFN Alfa-2a 180 mcg + Ribavirin 1200 mg | PEG-IFN Alfa-2a 180 mcg + Ribavirin 1600 mg | PEG-IFN Alfa-2a 270 mcg + Ribavirin 1200 mg | PEG-IFN Alfa-2a 270 mcg + Ribavirin 1600 mg
Number analyzed (Participants) | 46 | 47 | 47 | 47
log 10 copies/mL
  Baseline, (n=46,47,47,47) | 6.50 (0.45) | 6.61 (0.41) | 6.55 (0.44) | 6.53 (0.42)
  At Hour 72, (n=41,41,42,46) | 5.80 (0.54) | 5.82 (0.84) | 5.52 (0.67) | 5.49 (0.90)
  At Week 1, (n=44,47,45,46) | 5.74 (0.58) | 5.81 (0.92) | 5.42 (0.84) | 5.45 (0.97)
  At Week 2, (n=43,45,43,46) | 5.32 (0.91) | 5.37 (1.20) | 4.83 (1.12) | 4.84 (1.27)
  At Week 4, (n=44,45,44,46) | 4.35 (1.32) | 4.62 (1.38) | 3.94 (1.36) | 3.85 (1.41)
  At Week 12, (n=45,45,41,44) | 2.99 (1.55) | 3.10 (1.53) | 2.52 (1.28) | 2.75 (1.57)
  At Week 24, (n=42,45,40,37) | 2.76 (1.59) | 2.82 (1.58) | 2.25 (1.10) | 2.21 (1.32)

2. Secondary Outcome: Percentage of Participants With Sustained Virological Response
Description: SVR is defined as the percentage of participants with undetectable HCV RNA as measured by the Roche Amplicor HCV Test, v 2.0 (detection limit = 50 IU/ml) at the end of the 24-week untreated follow-up period.
Time Frame: Week 72
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PEG-IFN Alfa-2a 180 mcg + Ribavirin 1200 mg | PEG-IFN Alfa-2a 180 mcg + Ribavirin 1600 mg | PEG-IFN Alfa-2a 270 mcg + Ribavirin 1200 mg | PEG-IFN Alfa-2a 270 mcg + Ribavirin 1600 mg
Number analyzed (Participants) | 46 | 47 | 47 | 47
percentage of participants | 28.3 [15.25 to 41.27] | 31.9 [18.59 to 45.24] | 36.2 [22.43 to 49.91] | 46.8 [32.54 to 61.07]

3. Secondary Outcome: Percentage of Participants With Virological Response at the End of the Treatment Period
Description: Virological response at the end of the treatment period is defined as the percentage of participants with undetectable HCV RNA as measured by the Roche Amplicor HCV Test, v 2.0 (detection limit = 50 IU/mL) at the completion of the treatment period.
Time Frame: Week 48
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PEG-IFN Alfa-2a 180 mcg + Ribavirin 1200 mg | PEG-IFN Alfa-2a 180 mcg + Ribavirin 1600 mg | PEG-IFN Alfa-2a 270 mcg + Ribavirin 1200 mg | PEG-IFN Alfa-2a 270 mcg + Ribavirin 1600 mg
Number analyzed (Participants) | 46 | 47 | 47 | 47
percentage of participants | 45.7 [31.26 to 60.05] | 57.4 [43.31 to 71.58] | 55.3 [41.11 to 69.53] | 55.3 [41.11 to 69.53]

4. Secondary Outcome: Percentage of Participants With Virological Response At 12 Weeks After The End of The Treatment Period
Description: Virological response at 12 weeks after the end of the treatment period is defined as the percentage of participants with undetectable HCV RNA as measured by the Roche Amplicor HCV Test, v 2.0 (detection limit = 50 IU/mL) at 12 weeks after completion of the treatment period.
Time Frame: Week 60
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PEG-IFN Alfa-2a 180 mcg + Ribavirin 1200 mg | PEG-IFN Alfa-2a 180 mcg + Ribavirin 1600 mg | PEG-IFN Alfa-2a 270 mcg + Ribavirin 1200 mg | PEG-IFN Alfa-2a 270 mcg + Ribavirin 1600 mg
Number analyzed (Participants) | 46 | 47 | 47 | 47
percentage of participants | 28.3 [15.25 to 41.27] | 29.8 [16.71 to 42.86] | 34.0 [20.50 to 47.59] | 46.8 [32.54 to 61.07]

5. Secondary Outcome: Percentage of Participants With Adverse Events and Serious Adverse Events
Description: An adverse event (AE) is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events. A serious adverse event is any adverse event (SAE) that can result in death or is Life-threatening or required in-patient hospitalization or prolongation of existing hospitalization or results in persistent or significant disability/incapacity; or is a congenital anomaly/birth defect; or is medically significant or requires intervention to prevent one or other of the outcomes listed above.
Time Frame: Up to Week 72
Population: The safety population consisted of all participants who received at least one dose of either of the study drug and have at least one post-baseline safety assessment. Participants available at particular time point for assessment were included in the analysis.
  .
Measure: Number; unit: percentage of participants
Arm/Group | PEG-IFN Alfa-2a 180 mcg + Ribavirin 1200 mg | PEG-IFN Alfa-2a 180 mcg + Ribavirin 1600 mg | PEG-IFN Alfa-2a 270 mcg + Ribavirin 1200 mg | PEG-IFN Alfa-2a 270 mcg + Ribavirin 1600 mg
Number analyzed (Participants) | 46 | 47 | 47 | 47
percentage of participants
  Any AE | 100 | 100 | 100 | 100
  SAE | 9 | 13 | 13 | 11

6. Secondary Outcome: Percentage of Participants With Marked Laboratory Abnormalities
Description: Marked laboratory abnormalities are the values outside the roche defined reference range.It is hemoglobin 11.0 - 20.0 (g/dL),platelets 100 - 700 (10^9/L), lymphocyte 1.00 - 6.30 (10^9/L),neutrophils 1.50 or more (10^9/L), white blood cells(WBC) 3.0 - 18.0 (10^9/L),serum glutamic-pyruvic transaminase (SGPT) 0 - 60 (U/L), serum glutamic oxaloacetic transaminase (SGOT) 0 - 50 (U/L), alkaline phosphatase 0 - 190 (U/L),albumin was 27.0 or more (g/L),gamma glutamyl transferases (GGT) 0 - 120 (U/L),Total protein 55 - 87 (g/L),total bilirubin 0 - 34.2 (μmol/L),BUN 0 - 14.3 (mmol/L),creatinine 0 - 154 (μmol/L),chloride 95 - 115 (mmol/L),potassium 3.0 - 6.0 (mmol/L), sodium 130 - 150 (mmol/L),thyroid stimulating hormone (TSH) 0.0 - 10.0 (mU/L),triglycerides 0.00 - 2.83 (mmol/L), calcium 2.00 - 2.90 (mmol/L),phosphate 0.75 - 1.60 (mmol/L),Blood Glucose 2.80 - 11.10 (mmol/L),Uric Acid 0 - 600 (μmol/L),proteinuria 0 - 1 (0 to 4+), glycosuria 0 - 1 (0 to 4+), hematuria 0 - 1 (0 to 4+).
Time Frame: Up to Week 60
Population: The safety population consisted of all participants who received at least one dose of either of the study drug and have at least one post-baseline safety assessment. Participants available at particular time point for assessment where included in the analysis.
  .
Measure: Number; unit: percentage of participants
Groups:
- PEG-IFN Alfa-2a 180 mcg +Ribavirin 1200 mg: Participants received 180 mcg of PEG-IFN alfa-2a in 1 mL solution administered sc, once weekly + 1200 mg of ribavirin (200 mg/tablet) + ribavirin placebo (2 tablets) administered po daily in split doses for 48 weeks
Arm/Group | PEG-IFN Alfa-2a 180 mcg +Ribavirin 1200 mg | PEG-IFN Alfa-2a 180 mcg + Ribavirin 1600 mg | PEG-IFN Alfa-2a 270 mcg + Ribavirin 1200 mg | PEG-IFN Alfa-2a 270 mcg + Ribavirin 1600 mg
Number analyzed (Participants) | 45 | 47 | 46 | 47
percentage of participants
  Hematocrit (fraction) Low, (n=45,47,46,47) | 44 | 53 | 41 | 64
  Hemoglobin (g/dl) - Low, (n= 45,47,46,47) | 42 | 57 | 48 | 55
  Platelets Low, (n= 45,47,46,47) | 27 | 26 | 28 | 21
  WBC - High, [n= 45,47,46,47] | 0 | 2 | 0 | 0
  WBC - Low, (n= 45,47,46,47) | 76 | 72 | 70 | 74
  Lymphocytes High, (n= 45,47,46,47) | 0 | 0 | 0 | 2
  Lymphocytes Low (n= 45,47,46,47) | 73 | 68 | 72 | 72
  Neutrophils Low, (n= 45,47,46,47) | 82 | 79 | 74 | 74
  SGPT High, (n= 45,47,46,47) | 20 | 19 | 15 | 13
  Albumin Low, (n= 45,47,46,47) | 0 | 0 | 2 | 2
  Alkaline Phosphate High, (n= 45,47,46,47) | 0 | 0 | 2 | 0
  SGOT High, (n= 45,47,46,47) | 16 | 17 | 22 | 26
  GGT High, (n= 45,47,46,47) | 27 | 19 | 15 | 19
  Total Bilirubin High, (n= 45,47,46,47) | 9 | 6 | 2 | 2
  Total Protein High, (n= 45,47,46,47) | 0 | 0 | 0 | 4
  Bun High, (n= 45,47,46,47) | 0 | 2 | 0 | 0
  Chloride High, (n= 45,47,46,47) | 0 | 0 | 2 | 0
  Chloride Low (n= 45,47,46,47) | 0 | 2 | 0 | 2
  Creatinine High, (n= 45,47,46,47) | 0 | 2 | 0 | 0
  Potassium Low, (n= 45,47,46,47) | 0 | 2 | 0 | 0
  Sodium High, (n= 45,47,46,47) | 2 | 4 | 0 | 2
  Sodium Low, (n= 45,47,46,47) | 0 | 0 | 0 | 2
  TSH High, (n= 45,46,43,46) | 0 | 7 | 5 | 9
  Calcium Low, (n= 45,47,46,47) | 0 | 4 | 0 | 2
  Phosphate High, (n= 45,47,46,47) | 2 | 0 | 7 | 0
  Phosphate Low, (n= 45,47,46,47) | 31 | 36 | 20 | 30
  Random glucose High, (n= 45,47,46,47) | 2 | 11 | 4 | 6
  Triglycerides High, (n= 45,47,46,47) | 60 | 38 | 57 | 49
  Uric acid High (n= 45,47,46,47) | 9 | 11 | 2 | 15
  Glycosuria High, (n= 44,46,44,45) | 7 | 0 | 5 | 2
  Hematuria High, (n= 44,46,44,45) | 5 | 2 | 7 | 0
  Proteinuria High, (n= 44,46,44,45) | 2 | 2 | 5 | 0

7. Secondary Outcome: Percentage of Participants With Abnormal Vital Signs
Description: Vital signs (Systolic blood pressure, Diastolic blood pressure, Pulse rate) were considered to be abnormal and of potential clinical relevance if the values measured for these parameters represented a change from baseline of greater than 20% in the direction of worsening. High diastolic blood pressure is defined as >110 mmhg and >20% increase from baseline. High systolic blood pressure is defined as >180 mmhg and >20% increase from baseline. Low systolic blood pressure is defined as <85 mmhg and >20% decrease from baseline. High heart rate is defined as >120 beats/minute and >20% increase from baseline. Low heart rate is defined as < 50 beats/minute and >20% decrease from baseline.
Time Frame: Up to Week 72
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | PEG-IFN Alfa-2a 180 mcg + Ribavirin 1200 mg | PEG-IFN Alfa-2a 180 mcg + Ribavirin 1600 mg | PEG-IFN Alfa-2a 270 mcg + Ribavirin 1200 mg | PEG-IFN Alfa-2a 270 mcg + Ribavirin 1600 mg
Number analyzed (Participants) | 45 | 47 | 46 | 47
percentage of participants
  Diastolic BP, High (n=45,47,46,47) | 0 | 0 | 0 | 0
  Systolic BP High, (n=45,47,46,47) | 0 | 2 | 0 | 4
  Systolic BP Low, (n=45,47,46,47) | 0 | 0 | 2 | 0
  Heart Rate Low, (n=45,47,46,47) | 2 | 0 | 0 | 0
  Heart Rate, High, (n=45,47,46,47) | 0 | 0 | 0 | 0

8. Secondary Outcome: Total BDI-II (Beck Depression Inventory) Scores
Description: The BDI-II is a self-reported assessment of 21 items which included sadness, pessimism, past failure, loss of pleasure, guilty feelings, punishment feelings, self-dislike, self-criticalness, suicidal thoughts or wishes, crying, agitation, loss of interest, indecisiveness, worthlessness, loss of energy, changes in sleeping pattern, irritability, changes in appetite, concentration difficulty, tiredness or fatigue, loss of interest in sex that are summarized by treatment group. All except two items had four statements that were scored on a scale ranging from 0 to 3. The maximum total score was 63. The scores for each item were summed to obtain the total for that assessment. The participants neurological status could then be categorized as follows: minimal depression: 0 to 13; mild depression: 14 to 19; moderate depression: 20 to 28; and severe depression: 29 to 63. The BDI-II questionnaire was self-administered by the patient at each visit.
Time Frame: From Baseline (Day 1) to Week 72
Population: The safety population consisted of all participants who received at least one dose of either of the study drug and have at least one post-baseline safety assessment. Participants available at particular time point for assessment were included in the analysis.
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- PEG-IFN Alfa-2a 270 mcg+ Ribavirin 1600 mg: Participants received 270 mcg of PEG-IFN alfa-2a in 1-mL solution administered sc once weekly + 1600 mg of ribavirin (200 mg/tablet) administered po daily in split doses for 48 weeks
Arm/Group | PEG-IFN Alfa-2a 180 mcg + Ribavirin 1200 mg | PEG-IFN Alfa-2a 180 mcg + Ribavirin 1600 mg | PEG-IFN Alfa-2a 270 mcg + Ribavirin 1200 mg | PEG-IFN Alfa-2a 270 mcg+ Ribavirin 1600 mg
Number analyzed (Participants) | 46 | 47 | 47 | 47
Units on a scale
  Baseline, n=46,46,47,46 | 3.52 (4.34) | 4.39 (4.82) | 4.23 (4.31) | 4.43 (4.70)
  Week 1, (n=43,44,43,45) | 4.24 (4.53) | 4.45 (4.33) | 4.81 (4.40) | 3.96 (3.76)
  Week 2, (n=43,44,43,47) | 4.84 (4.51) | 4.71 (5.16) | 5.60 (5.31) | 5.22 (5.27)
  Week 4, (n=42,45,44,45) | 6.31 (6.03) | 5.79 (5.50) | 7.21 (7.51) | 6.07 (4.77)
  Week 6, (n=41,41,43,44) | 6.32 (6.33) | 6.49 (5.40) | 8.19 (7.42) | 6.64 (5.71)
  Week 8, (n=38,42,42,40) | 6.20 (6.06) | 6.24 (5.39) | 8.02 (7.16) | 7.69 (6.90)
  Week 12, (n=44,46,42,44) | 6.82 (6.93) | 7.09 (5.76) | 8.09 (7.19) | 8.09 (8.12)
  Week 18, (n=43,44,42,40) | 8.04 (7.46) | 8.31 (6.91) | 8.62 (6.96) | 8.13 (7.86)
  Week 24, (n=43,45,41,37) | 7.07 (7.17) | 7.43 (7.04) | 8.80 (7.79) | 8.05 (6.37)
  Week 30, (n=38,42,39,34) | 8.03 (7.98) | 7.89 (6.80) | 9.35 (8.07) | 7.74 (6.14)
  Week 36, (n=36,42,37,33) | 7.50 (7.13) | 8.63 (8.09) | 7.82 (7.48) | 9.45 (8.71)
  Week 42, (n=35,37,35,32) | 7.49 (7.22) | 8.33 (8.06) | 8.00 (5.50) | 8.13 (5.43)
  Week 48, (n=34,40,31,29) | 7.48 (7.79) | 7.89 (7.79) | 7.92 (5.00) | 7.93 (5.13)
  Week 52, (n=31,36,32,28) | 4.56 (6.87) | 6.62 (8.59) | 4.22 (4.47) | 4.21 (3.79)
  Week 60, (n=34,34,31,28) | 4.47 (6.18) | 5.18 (6.61) | 3.40 (4.08) | 3.12 (4.00)
  Week 72, (n=28,37,28,29) | 5.00 (7.69) | 5.14 (6.61) | 2.92 (4.48) | 2.80 (4.59)

9. Primary Outcome: Percentage of Participants With Virological Response Over Time to Week 24
Description: Virological response over time to Week 24 is defined as the percentage of participants with undetectable HCV RNA as measured by the Roche Amplicor HCV Test, V. 2.0 (detection limit = 50 IU/mL) at 72 hours and at weeks 1, 2, 12, and 24.
Time Frame: 72 hours post-dose, Weeks 1, 2, 4, 12, and 24
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PEG-IFN Alfa-2a 180 mcg +Ribavirin 1200 mg | PEG-IFN Alfa-2a 180 mcg + Ribavirin 1600 mg | PEG-IFN Alfa-2a 270 mcg + Ribavirin 1200 mg | PEG-IFN Alfa-2a 270 mcg + Ribavirin 1600 mg
Number analyzed (Participants) | 46 | 47 | 47 | 47
percentage of participants
  At Hour 72 | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00]
  At Week 1 | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00]
  At Week 2 | 0.00 [0.00 to 0.00] | 2.1 [0.00 to 6.25] | 2.1 [0.00 to 6.25] | 2.1 [0.00 to 6.25]
  At Week 4 | 2.2 [0.00 to 6.39] | 8.5 [0.53 to 16.49] | 10.6 [1.82 to 19.45] | 12.8 [3.23 to 22.31]
  At Week 12 | 47.8 [33.39 to 62.26] | 38.3 [24.40 to 52.20] | 53.2 [38.93 to 67.46] | 51.1 [36.77 to 65.36]
  At Week 24 | 56.5 [42.20 to 70.85] | 55.3 [41.11 to 69.53] | 59.6 [45.54 to 73.60] | 68.1 [54.76 to 81.41]

10. Primary Outcome: Percentage of Participants With Predicted Sustained Virological Response
Description: The predicted sustained virological response (SVR) for each treatment group, is determined using a model based on the log10-transformed HCV viral load in copies/mL at Week 4 and the virological response status at Week 12. Each participant was classified as a predicted SVR if p was ≥ 0.5 or as a non-SVR if p was <0.5. The percentage was calculated from the number of participant (N) analyzed under "Distribution of the predicted probability of an SVR."
Time Frame: Week 4 and 12
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | PEG-IFN Alfa-2a 180 mcg + Ribavirin 1200 mg | PEG-IFN Alfa-2a 180 mcg + Ribavirin 1600 mg | PEG-IFN Alfa-2a 270 mcg + Ribavirin 1200 mg | PEG-IFN Alfa-2a 270 mcg + Ribavirin 1600 mg
Number analyzed (Participants) | 44 | 45 | 44 | 46
percentage of participants | 40.9 | 31.1 | 47.7 | 50.0

ADVERSE EVENTS:
Time Frame: Up to Week 72
Description: Serious adverse events and non-serious adverse events are reported in Safety Analysis Set, which consists of all participants who received at least one dose of study medication and had a safety assessment performed post-baseline.
Groups:
- PEG-IFN Alfa-2a 180 mcg +Ribavirin 1200 mg: Participants received 180 mcg of PEG-IFN alfa-2a in 1-ml solution administered [subcutaneously] sc, once in a week + 1200 mg of ribavirin (200 mg/tablet) + ribavirin placebo (2 tablets) administered [orally ] po daily in split doses for 48 weeks
- PEG-IFN Alfa-2a 180 mcg + Ribavirin 1600 mg: Participants received 180 mcg of PEG-IFN alfa-2a in 1-ml solution administered sc once in a week + 1600 mg of ribavirin (200 mg/tablet) administered po daily in split doses for 48 weeks.
- PEG-IFN Alfa-2a 270 mcg + Ribavirin 1200 mg: Participants received 270 mcg of PEG-IFN alfa-2a in 1-ml solution administered sc once in a week + 1200 mg of ribavirin (200 mg/tablet) + ribavirin placebo (2 tablets) administered po daily in split doses for 48 weeks
- PEG-IFN Alfa-2a 270 mcg + Ribavirin 1600 mg: Participants received 270 mcg of PEG-IFN alfa-2a in 1-ml solution administered sc once in a week + 1600 mg of ribavirin (200 mg/tablet) administered po daily in split doses for 48 weeks.
Arm/Group | PEG-IFN Alfa-2a 180 mcg +Ribavirin 1200 mg | PEG-IFN Alfa-2a 180 mcg + Ribavirin 1600 mg | PEG-IFN Alfa-2a 270 mcg + Ribavirin 1200 mg | PEG-IFN Alfa-2a 270 mcg + Ribavirin 1600 mg
Serious Adverse Events (participants affected / at risk) | 4/46 | 6/47 | 6/47 | 5/47
Other Adverse Events (participants affected / at risk) | 46/46 | 46/47 | 47/47 | 47/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PEG-IFN Alfa-2a 180 mcg +Ribavirin 1200 mg (N=46) | PEG-IFN Alfa-2a 180 mcg + Ribavirin 1600 mg (N=47) | PEG-IFN Alfa-2a 270 mcg + Ribavirin 1200 mg (N=47) | PEG-IFN Alfa-2a 270 mcg + Ribavirin 1600 mg (N=47)
Pneumonia (Infections and infestations) | 0 | 0 | 2 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 1
Staphylococcal Sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 1
Anaemia Haemolytic Autoimmune (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0
Homicidal Ideation (Psychiatric disorders) | 0 | 0 | 0 | 1
Psychotic disorder (Psychiatric disorders) | 1 | 0 | 0 | 0
Suicidal Ideation (Psychiatric disorders) | 0 | 0 | 0 | 1
Suicide attempt (Psychiatric disorders) | 1 | 0 | 0 | 0
Ankle Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Road Traffic Accident (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Non Hodgkin's Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Retinal Vascular Disorder (Eye disorders) | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 1 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Sarcoidosis (Immune system disorders) | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Haemorrhagic Ovarian Cyst (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Thrombosis (Vascular disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PEG-IFN Alfa-2a 180 mcg +Ribavirin 1200 mg (N=46) | PEG-IFN Alfa-2a 180 mcg + Ribavirin 1600 mg (N=47) | PEG-IFN Alfa-2a 270 mcg + Ribavirin 1200 mg (N=47) | PEG-IFN Alfa-2a 270 mcg + Ribavirin 1600 mg (N=47)
Anaemia (Blood and lymphatic system disorders) | 3 | 6 | 4 | 12
Vertigio (Ear and labyrinth disorders) | 0 | 0 | 3 | 1
Vision blurred (Eye disorders) | 5 | 3 | 5 | 3
Abdominal Pain (Gastrointestinal disorders) | 0 | 4 | 2 | 3
Abdominal pain upper (Gastrointestinal disorders) | 4 | 3 | 6 | 4
Constipation (Gastrointestinal disorders) | 3 | 2 | 4 | 3
Diarrhoea (Gastrointestinal disorders) | 12 | 9 | 11 | 10
Dry Mouth (Gastrointestinal disorders) | 2 | 4 | 6 | 3
Dyspepsia (Gastrointestinal disorders) | 3 | 4 | 4 | 5
Nausea (Gastrointestinal disorders) | 18 | 20 | 18 | 18
Stomatitis (Gastrointestinal disorders) | 1 | 4 | 1 | 1
Toothache (Gastrointestinal disorders) | 4 | 3 | 1 | 4
Vomiting (Gastrointestinal disorders) | 6 | 5 | 7 | 5
Asthenia (General disorders) | 3 | 4 | 2 | 5
Chest discomfort (General disorders) | 0 | 3 | 0 | 3
Chills (General disorders) | 15 | 14 | 19 | 17
Fatigue (General disorders) | 36 | 32 | 35 | 34
Injection site erythema (General disorders) | 10 | 9 | 6 | 5
Injection site rash (General disorders) | 2 | 3 | 0 | 1
Injection site reaction (General disorders) | 4 | 3 | 2 | 1
Irritability (General disorders) | 14 | 14 | 12 | 16
Malaise (General disorders) | 1 | 3 | 5 | 3
Pain (General disorders) | 4 | 1 | 2 | 2
Pyrexia (General disorders) | 12 | 14 | 16 | 14
Cellulitis (Infections and infestations) | 2 | 1 | 4 | 0
Herpes Simplex (Infections and infestations) | 3 | 1 | 2 | 1
Oral Candidiasis (Infections and infestations) | 1 | 3 | 0 | 0
Sinusitis (Infections and infestations) | 3 | 2 | 2 | 2
Tooth infection (Infections and infestations) | 0 | 3 | 0 | 0
Upper Respiratory tract infection (Infections and infestations) | 2 | 5 | 3 | 6
Urinary tract infection (Infections and infestations) | 0 | 1 | 4 | 0
Contusion (Injury, poisoning and procedural complications) | 3 | 1 | 2 | 1
Weight Decreased (Investigations) | 6 | 4 | 5 | 7
Anorexia (Metabolism and nutrition disorders) | 6 | 4 | 6 | 4
Decreased Appetite (Metabolism and nutrition disorders) | 5 | 5 | 9 | 8
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 2 | 0 | 5 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 13 | 16 | 16 | 15
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 11 | 4 | 3
Muscle spasm (Musculoskeletal and connective tissue disorders) | 2 | 5 | 3 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 14 | 15 | 19 | 16
Disturbance in attention (Nervous system disorders) | 9 | 4 | 7 | 6
Dizziness (Nervous system disorders) | 12 | 9 | 7 | 9
Dysgeusia (Nervous system disorders) | 3 | 0 | 8 | 4
Headache (Nervous system disorders) | 24 | 18 | 22 | 21
Memory impairment (Nervous system disorders) | 8 | 5 | 3 | 4
Tremor (Nervous system disorders) | 1 | 2 | 4 | 0
Anger (Psychiatric disorders) | 3 | 1 | 1 | 0
Anxiety (Psychiatric disorders) | 7 | 3 | 7 | 8
Depression (Psychiatric disorders) | 14 | 20 | 11 | 16
Insomnia (Psychiatric disorders) | 18 | 20 | 22 | 24
Mood altered (Psychiatric disorders) | 0 | 1 | 4 | 0
Sleep disorder (Psychiatric disorders) | 3 | 3 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 12 | 12 | 8
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 | 12 | 8 | 12
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 6 | 1 | 5 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 3 | 1
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 4 | 2
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 3 | 1
Respiratory tract conjestion (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 3 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 4 | 5 | 5 | 6
Dry Skin (Skin and subcutaneous tissue disorders) | 3 | 3 | 4 | 5
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 5 | 1 | 2 | 8
Night Sweats (Skin and subcutaneous tissue disorders) | 2 | 1 | 3 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 7 | 3 | 6 | 3
Rash (Skin and subcutaneous tissue disorders) | 12 | 11 | 15 | 12
Rash Generalised (Skin and subcutaneous tissue disorders) | 2 | 2 | 2 | 4
Hypertension (Vascular disorders) | 0 | 0 | 1 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.